CLINICAL TRIAL: NCT05278910
Title: Innovative Methods to Reduce Emissions and Health Impacts of Deep-frying
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Academia Sinica, Taiwan (Other)
Responsible Party: Principal Investigator, Wen-Harn Pan, Distinguished Research Fellow, Principal Investigator, Academia Sinica, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AS-IRB01-21006
Record Dates: First submitted 2022-01-16; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Soybean Oil; Fish Oils; Vegetables

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Soybean oil + Roasted wheat flour (Placebo Comparator): Assign soybean oil capsule and roasted wheat flour.
  Interventions: Other: Soybean oil + Roasted wheat flour
- Fish oil + Roasted wheat flour (Experimental): Assign fish oil capsule and roasted wheat flour.
  Interventions: Dietary Supplement: Fish oil + Roasted wheat flour
- Soybean oil + Vegetable and fruit extracts (Experimental): Assign soybean oil capsule and Vegetable and fruit extracts.
  Interventions: Dietary Supplement: Soybean oil + Vegetable and fruit extracts
- Fish oil + Vegetable and fruit extracts (Experimental): Assign fish oil capsule and Vegetable and fruit extracts.
  Interventions: Dietary Supplement: Fish oil + Vegetable and fruit extracts

INTERVENTIONS:
Other: Soybean oil + Roasted wheat flour — Assign soybean oil capsule and roasted wheat flour
  Arms: Soybean oil + Roasted wheat flour
Dietary Supplement: Fish oil + Roasted wheat flour — Assign fish oil and roasted wheat flour
  Arms: Fish oil + Roasted wheat flour
Dietary Supplement: Soybean oil + Vegetable and fruit extracts — Assign soybean oil and vegetable and fruit extracts
  Arms: Soybean oil + Vegetable and fruit extracts
Dietary Supplement: Fish oil + Vegetable and fruit extracts — Assign fish oil and vegetable and fruit extracts
  Arms: Fish oil + Vegetable and fruit extracts

SUMMARY:
Cooking oil fume (COF) is a significant source of PM2.5 for poorly ventilated space indoors and in urban streets near restaurants or night markets. Modern Chinese cooking produces high concentration of COF especially from deep-frying foods and stirred frying. Emission from high-temperature frying has been classified by the IARC as Group 2A carcinogen. Cooks are at high risk of exposure to toxic compounds from cooking fumes. However, more of the COF-related studies focused on the home kitchen and less addresses the problems in the restaurants. Studying health hazards and biomarkers of cooks may provide opportunities to understand biological mechanisms and to search and test efficacy for measures to overturn such risks.

The investigators will recruit 80 cooks who handle deep-frying and stirred frying on daily basis. The 80 cooks will be randomized to 4 groups: (1) control, (2) vegetable and fruits extract (V&F) group, (3) fish oil group, and (4) V&F-fish oil group will be provided to the participants for 2 months V&F capsules (equivalent to 4 servings a day) and fish oil capsules (1~1.5 serving a day) and placebos of the same appearance. Heart rate variability (HRV), pulmonary functions, bio-markers, oxylipins and metabolomics profile will be measured as outcomes.

ELIGIBILITY:
Exclusion Criteria:

1. Acute diseases in the past 2 weeks
2. Taking anti-oxidant supplements in the past month
3. Taking steroid or non-steroidal anti-inflammatory drugs (such as Aspirin and Panadol) in the past week
4. Under hormone replacement therapy
5. Cancer and other severe diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-14 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HRV | baseline and 2 months later
  Change in heart rate variability (HRV)
Change in pulmonary functions (TLC) | baseline and 2 months later
  Change in TLC in L
Change in pulmonary functions (FVC) | baseline and 2 months later
  Change in FVC in L
Change in pulmonary functions (FEV1) | baseline and 2 months later
  Change in FEV1 in L
Change in pulmonary functions (PEF) | baseline and 2 months later
  Change in PEF in L/sec
Change in pulmonary functions (FEF) | baseline and 2 months later
  Change in FEF in L/sec
Change in oxidative stress marker | baseline and 2 months later
  Change in urinary 8-OHdG for DNA damage
Change from baseline in concentrations of inflammatory markers | baseline and 2 months later
  Inflammatory markers include IL-1β, IL-2, IL-4, IL-6, IL-10, IL-12, IL-13, IL-17A, IL-23, IL-33, TNF- α, IFN-γ, CXCL1, CXCL9, and CXCL10 (IP-10) in blood

SECONDARY OUTCOMES:
Change in blood cell count | baseline and 2 months later
  Blood cell count is measured by Completed Blood Count Test
Change in blood cholesterol markers | baseline and 2 months later
  Blood cholesterol markers include HDL in mg/dL, LDL in mg/dL, TG in mg/dL and total cholesterol in mg/dL
Change in blood sugar (HbA1C) | baseline and 2 months later
  Change in HbA1C in %
Change in blood sugar (glucose) | baseline and 2 months later
  Change in glucose in mg/dL
Change in liver function | baseline and 2 months later
  The markers of liver function include GOT in U/L and GPT in U/L
Change in kidney function | baseline and 2 months later
  The markers of kidney function include creatinine in mg/dL, uric acid in mg/dL, BUN in mg/dL, microalbumin in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Harn Pan, PhD, Principal Investigator — Institute of Biomedical Sciences, Academia Sinica